CLINICAL TRIAL: NCT02232022
Title: Occult Paroxysmal Atrial Fibrillation in Non-Cryptogenic Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Jeffrey Katz, Chief, Vascular Neurology, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-336
Record Dates: First submitted 2014-09-02; First posted 2014-09-04 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-06

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Ischemic stroke; Atrial fibrillation; Insertable cardiac monitor; Non-cryptogenic
MeSH Terms: conditions — Ischemic Stroke; Stroke; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NonCryptogenic Ischemic Stroke Patients (Experimental): Patients with non-cryptogenic ischemic stroke will be enrolled within 10 days of stroke onset
  Interventions: Device: Reveal LINQ Insertable Cardiac Monitor

INTERVENTIONS:
Device: Reveal LINQ Insertable Cardiac Monitor

SUMMARY:
The purpose of this study is to determine the incidence of paroxysmal atrial fibrillation (AF) in ischemic stroke patients who have a presumed known stroke etiology other than atrial fibrillation.

DETAILED DESCRIPTION:
Recent studies suggest that their is a relatively high incidence of silent paroxysmal atrial fibrillation (PAF) in cryptogenic ischemic stroke patients. Detection of silent PAF in this population, however, requires prolonged cardiac monitoring. On the other hand, there is no understanding of the frequency of silent PAF in patients with a "known" or presumed etiology for their ischemic stroke other than AF. If this incidence is also found to be significant, a dramatic change in stroke evaluation and management would likely occur. This study intends to find the incidence of PAF in a population of recent (within 7 days) ischemic stroke patients (or MRI positive "transient ischemic attack (TIA)" patients) who have presumed etiology for their stroke other than atrial fibrillation or other high risk cardiac lesion. Stroke etiology will be determined through a standard post-stroke evaluation that includes:

* Brain MRI
* 12-lead electrocardiogram (ECG) for AF detection
* 24-h ECG monitoring for AF detection (eg, Holter monitor or cardiac telemetry)
* Transthoracic and/or Transesophageal echocardiogram
* CT or MR angiography of the head and neck
* Hypercoagulable blood panel for patients less than 55 years-old. Preliminary hypercoagulable work-up within 7 days will include the antiphospholipid antibody syndrome results, which will be needed to determine stroke management. All other results, which could take longer to return, including genetic tests of hypercoagulability, rarely change stroke management.

To find occult PAF in this population, participants will have an insertable cardiac monitor (Reveal LINQ ICM) implanted within 7 days of the incident stroke and will be monitored for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a recent ischemic stroke or transient ischemic attack (TIA) with brain infarction on brain imaging.
* No history of atrial fibrillation or finding of atrial fibrillation on standard inpatient monitoring (electrocardiogram, telemetry, 24-hour Holter monitor)
* Have a presumed stroke etiology: Lacunar or small vessel thrombosis, extra-cranial or intracranial atherosclerotic stenosis or dissection, arteriopathy or vasculitis, hypercoagulable state, aortic arch plaque with or without mobile elements, or evidence of a low-risk cardiac source (e.g., patent foramen ovale with or without atrial septal aneurysm and with or without evidence of venous thromboembolic source).
* Have virtual CHADS2 score ≥3 or
* Have 2 or more of the following co-morbidities: obstructive sleep apnea, coronary artery disease, (Chronic Pulmonary Obstructive Disease (COPD), hyperthyroidism, Body Mass Index> 30, prior myocardial infarction, prolonged PR interval (>175 ms) or renal impairment (GFR 30-60).
* Patient or legally authorized representative who is willing to sign written consent form.
* Patient is ≥40 years old (patients younger than 40 years old have a very low likelihood of having atrial fibrillation and are therefore excluded from the study).
* Patient can have the device implanted within 7 days of the incident ischemic event

Exclusion Criteria:

* Documented history of AF or atrial flutter.
* Evidence of a high-risk cardiac source of embolism (Left Ventricular or Left Atrial thrombus or "smoke," emboligenic valvular lesion or tumor)
* Untreated hyperthyroidism.
* Myocardial infarction or coronary bypass grafting within 1 month prior to the stroke/TIA.
* Valvular disease requiring immediate surgical intervention.
* Permanent indication for anticoagulation at enrollment.
* Permanent oral anticoagulation contraindication.
* Already included in another clinical trial that will affect the objectives of this study.
* Life expectancy is less than 1 year.
* Pregnancy. Urine or serum pregnancy test is required for women of child bearing potential to exclude pregnancy.
* Patient is indicated for implant with a pacemaker, implantable cardioverter-defibrillator, CRT device, or an implantable hemodynamic monitoring system
* Patient is not fit, or is unable or unwilling to follow the required procedures of the Clinical Investigation Plan.
* Cryptogenic Stroke: A stroke/TIA will be considered cryptogenic if no cause is determined despite extensive inpatient workup according to the standard diagnostic protocol at North Shore University Hospital.

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Katz, MD, Principal Investigator — Northwell Health
Locations (2):
- United States (2):
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NonCryptogenic Ischemic Stroke Patients: In this pilot prospective cohort study of non-CIS patients from September 2014 to September 2017. Patients were implanted within 10 days of stroke onset with the Reveal LINQ insertable cardiac monitor and monitored until PAF detection or a minimum of 12 months. Inclusion required diagnosis of a non-AF stroke etiology, age≥40, and either a virtual CHADS2 score ≥3 or ≥2 PAF related comorbidities.
Period: Overall Study
Arm/Group | NonCryptogenic Ischemic Stroke Patients
Started | 53
Completed | 51
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- NonCryptogenic Ischemic Stroke Patients: In this pilot prospective cohort study of non-CIS patients from September 2014 to September 2017, 53 patients were enrolled. 51/53 patients were implanted within 10 days of stroke onset with the Reveal LINQ insertable cardiac monitor and monitored until PAF detection or a minimum of 12 months.
  Inclusion required diagnosis of a non-AF stroke etiology, age≥40, and either a virtual CHADS2 score ≥3 or ≥2 PAF related comorbidities.
Arm/Group | NonCryptogenic Ischemic Stroke Patients
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 32
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 53
Baseline AF Assessment [Count of Participants; unit: Participants] — Baseline AF Assessment completed using 24 hour ECG monitoring
  Participants | 53

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Paroxysmal Atrial Fibrillation (AF) in Ischemic Stroke Patients
Description: The incidence of paroxysmal atrial fibrillation (AF) in ischemic stroke patients who have a presumed known stroke etiology other than atrial fibrillation.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- NonCryptogenic Ischemic Stroke: Reveal LINQ Insertable Cardiac Monitor
Arm/Group | NonCryptogenic Ischemic Stroke
Number analyzed (Participants) | 51
Participants | 6

2. Secondary Outcome: Patients Who Are Diagnosed With AF Who Are Changed to Anticoagulant Therapy.
Description: Percentage of patients who are diagnosed with AF who are changed to anticoagulant therapy.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | NonCryptogenic Ischemic Stroke Patients
Number analyzed (Participants) | 6
Participants | 5

3. Secondary Outcome: Duration of AF Episodes.
Description: Duration of AF episodes (mean and range).
Time Frame: 1 year
Measure: Mean (Full Range); unit: min
Arm/Group | NonCryptogenic Ischemic Stroke Patients
Number analyzed (Participants) | 6
min | 237 [1 to 1122]

4. Secondary Outcome: Percentage of Asymptomatic AF
Description: Percentage of asymptomatic AF episodes.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- NonCryptogenic Ischemic Stroke Patients: Reveal LINQ Insertable Cardiac Monitor.
Arm/Group | NonCryptogenic Ischemic Stroke Patients
Number analyzed (Participants) | 6
Participants | 6

5. Secondary Outcome: Incidence of Recurrent Stroke
Description: Incidence of recurrent ischemic stroke.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | NonCryptogenic Ischemic Stroke Patients
Number analyzed (Participants) | 53
Participants | 2

6. Secondary Outcome: Number of Patients That Had Multiple AF Episodes
Description: Number of patients that had multiple AF episodes.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | NonCryptogenic Ischemic Stroke
Number analyzed (Participants) | 6
Participants | 4

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | NonCryptogenic Ischemic Stroke Patients
All-Cause Mortality (participants affected / at risk) | 1/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 1/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NonCryptogenic Ischemic Stroke Patients (N=51)
Device Erosion (Skin and subcutaneous tissue disorders) | 1 — 1 patient had a complication of impending device erosion through the skin. Managed with antibiotics and device removal.

LIMITATIONS AND CAVEATS:
Relatively small sample size limits our study's power to detect and confirm all factors associated with PAF detection. The number of non-PAF patients lost to follow-up by 6 and 12 months that may have resulted in an underestimation of PAF burden.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT02232022/Prot_SAP_000.pdf